CLINICAL TRIAL: NCT04903002
Title: Evaluating the Efficacy of Intranasal Oxytocin on Pain and Function Among Individuals Who Experience Chronic Pain: a Multisite, Placebo-controlled, Blinded, Sequential, Within-subjects Crossover Trial
Brief Title: Evaluating the Efficacy of Intranasal Oxytocin on Chronic Pain
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: University of Calgary (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIHR-PG#426528
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a triple-blind study. In order to protect against expectation effects and biases, neither site investigators nor patients will know which nasal spray contains oxytocin or which sequence of conditions patients are assigned. The allocation sequence will be concealed from researchers using automated randomization. The bottles containing 24-IU oxytocin, 48-IU oxytocin, and placebo will be identical in appearance, smell, texture and taste, and only identifiable through a color labeling system known to the site pharmacists and study sponsor. Each site's randomization sequence will be accessed by the site pharmacist and bottles prepared accordingly. The RA assessing outcomes will be unaware of condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crossover sequence 1: Oxytocin first (Other): Patients receive 2-weeks courses of 24-IU oxytocin, placebo, 48-IU oxytocin.
  Interventions: Drug: 24-IU oxytocin; Drug: 48-IU oxytocin; Drug: Placebo
- Crossover sequence 2: placebo first (Other): Patients receive 2-weeks courses of placebo, 24-IU oxytocin, 48-IU oxytocin.
  Interventions: Drug: 24-IU oxytocin; Drug: 48-IU oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: 24-IU oxytocin — Patients will self-administer a 2-week course of 24-IU intranasal oxytocin [4-IU per puff (12-IU delivered to each nostril); Syntocinon, Novartis, Switzerland], twice per day (once in the morning and once in the evening).
Drug: 48-IU oxytocin — Patients will self-administer a 2-week course of 48-IU intranasal oxytocin [4-IU per puff (24-IU delivered to each nostril); Syntocinon, Novartis, Switzerland], twice per day (once in the morning and once in the evening).
Drug: Placebo — Patients will receive an intranasal placebo containing the same ingredients as the oxytocin nasal spray with the exception of active oxytocin. Administration schedule and procedure will be identical to that described in 24-IU oxytocin.

SUMMARY:
One in five Canadians live with chronic pain, defined as pain that lasts longer than 3-months. Living with chronic pain has a detrimental impact on physical health, emotional health, and quality of life. Current treatments rarely result in pain relief and often do not meaningfully improve physical or emotional function. Further, medication used to treat pain often causes unwanted symptoms. There is a need to develop new treatments to help manage chronic pain. The use of a nasal spray containing manufactured oxytocin may improve pain management. Oxytocin is produced in the human body and has been shown to impact the pain pathway in animals. Our project tests whether the use of a nasal spray containing oxytocin will improve pain and function in men and women who live with chronic pain. Men and women with chronic nerve, muscle, or pelvic pain will be recruited in Vancouver, Calgary, and St. John's. Each person will be assigned to complete three interventions in a random order. Each intervention involves using a nasal spray twice per day over a 2-week period. The nasal spray will contain a small dose of oxytocin during one intervention and a medium dose during the second intervention. The nasal spray during the final intervention will have no oxytocin. This final intervention is a control intervention that will allow us to measure the effect of simply taking a nasal spray (i.e., the impact of expectation). Participants and researchers will not know which interventions involve the use of oxytocin. Participants will rate their pain and function each day throughout each task. The investigators will calculate each person's score on pain and function. The investigators will test whether participants report less pain and better function when they use oxytocin compared to the control. The results of this project may improve pain, function, and quality of life among those who live with chronic pain.

DETAILED DESCRIPTION:
Background and Importance: Chronic pain affects 1 in 5 Canadians and is associated with considerable burden, both individual (disability, reduced physical and emotional function) and economic ($43 billion annual cost to the economy). Available treatments for chronic pain rarely resolve symptoms, may be associated with addiction and often do not improve function. There is a need for analgesics that are non-addictive, have low adverse effect profiles, and offer effective relief.

Our work suggests that oxytocin (OT), a neuropeptide produced in the hypothalamus, may be a safe and effective adjuvant analgesic for a broad patient population. There are three mechanisms through which OT may decrease pain sensitivity: 1) a direct hypothalamo-spinal projection transports OT to the dorsal horn, reducing pain signaling from the periphery to the brain; 2) binding to opioid receptors and stimulating endogenous opioid release in the brain; and 3) improving mood, anxiety, and stress. Our team published a systematic review of the effect of OT on pain showing that 29/33 animal investigations report that OT decreases pain. It is difficult to draw firm conclusions about the effect of OT on pain in humans due to a paucity of methodologically rigorous trials.

Goals / Research Aim: To evaluate the efficacy of intranasal OT as an adjuvant treatment to improve pain and function among men and women with chronic pain.

Methods:

Design: Multi-site, dose-response, placebo-controlled, blinded, sequential, within-subjects crossover trial.

Outcomes: As recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials, the primary outcome is change in pain-intensity assessed using the Brief Pain Inventory obtained from daily diaries.

Conditions: Experimental 1: 2-week course of 24-IU intranasal OT administered twice daily. Experimental 2: 2-week course of 48-IU intranasal OT administered twice daily. Control: 2-week course of intranasal placebo. Wash-Out: 2-week period occurring between each condition to allow OT to clear the system.

Recruitment: Patients with chronic neuropathic, musculoskeletal and pelvic pain will be recruited from 3 sites: Vancouver, Calgary, and St. John's. Patients will be randomized to one of 2 sequences (24-IU OT, placebo, 48-IU OT; placebo, 24-IU OT; 48-IU OT). Randomization will be centralized and stratified by site.

Blinding: Patients, researchers, and outcome assessors will be blind to condition.

Sample Size: 336 patients (112 per site) are required to detect a clinically significant (1-point; d = .50) change in pain using covariate adjusted repeated measures design with alpha = .05, power = .80, and one cluster (site).

Expected Outcomes: Provide a definitive answer regarding the efficacy of OT to improve pain and function in chronic pain in humans. An efficacy trial of this nature is a necessary prerequisite to conducting a translation trial which is aimed at improving the uptake and utilization of proven therapies in clinical practice and community settings.

ELIGIBILITY:
Inter-Site Inclusion Criteria:

1. Adult (> 18 years) men and premenopausal women;
2. On stable medication for pain management for 3 months or more with no anticipated changes during the 10-weeks of this trial;
3. Moderate pain at baseline (i.e., a score of 4-8 on a 10-point numeric rating scale) to prevent floor and ceiling effects.
4. Can commit the use of two forms of effective contraception (e.g., barrier methods), or one highly effective method, including abstinence, intrauterine device, intrauterine system (IUS), vasectomy, tubal ligation, or hormonal contraceptive (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants)

Intra-Site Inclusion Criteria:

1. Surrey, BC: Men and women with primary neuropathic pain - pain arising as a direct consequence of a lesion or disease affecting the central or peripheral nervous system - will be eligible. Neuropathic pain will be screened for using a score of 3+ on the Douleur Neuropathique 4 Interview, and confirmed through investigation (e.g., electromyography).
2. Calgary, AB: Women with chronic (intermittent or constant) pelvic musculoskeletal pain (i.e., located primarily in the pelvic region and reproducible on palpation of the pelvic floor) who have not received a hysterectomy will be eligible. Women with a primary diagnosis of endometriosis, dysmenorrhea, functional bowel disorder, interstitial cystitis, fibromyalgia or sacroiliac instability as defined by European Guidelines, will be excluded.
3. Carbonear NL: Men and women with primary musculoskeletal pain of back, neck, or shoulder origin will be eligible. Pain will be assessed using the BPI-SF and confirmed through physical examination.

Exclusion Criteria:

1. Positive urine pregnancy test or contemplating pregnancy;
2. Concurrent use of another nasal spray;
3. Nasal pathology (e.g., ears, nose, and throat diagnosis);
4. Diabetes insipidus;
5. Current diagnosis or history of cancer
6. Significant unmanaged psychopathology (e.g., severe depression as indicated by a score ≥ 15 on the Patient Health Questionnaire -9) due to its inverse association with patient adherence to procedures; and
7. Receiving hormone treatment for gender-related motivations.
8. documented cardiovascular event (e.g., myocardial infarction)
9. known prolongation of the QTc interval; 10) known hypersensitivity to oxytocin
10. known latex allergy
11. known or suspected renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Change from Day 1 to Day 14 of nasal spray administration.
  Pain severity index on the Brief Pain Inventory - Short Form (BPI-SF). Mean scores range from 0 to 10 with higher scores indicating greater pain.
Pain-related interference | Change from Day 1 to Day 14 of nasal spray administration.
  Pain interference index on the Brief Pain Inventory - Short Form (BPI-SF). Mean scores range from 0 to 10 with higher scores indicating greater pain-related interference.

SECONDARY OUTCOMES:
Emotional function | Change from Day 1 to Day 14 of nasal spray administration.
  Depression, Anxiety and Stress scale (DASS). Scores are calculated for 3 subscales that are each composed of 7-items (Depression, Anxiety and Stress). Scores on subscales range between 0 and 21 with higher scores reflecting greater reports of Depression, Anxiety or Stress.
Sleep Disturbance | Change from Day 1 to Day 14 of nasal spray administration.
  Sleep problems index on the Medical Outcomes Study Sleep Scale
Global Impression of Change | Rated at Day 14 of nasal spray administration
  Patient Global Impression of Change Scale (PGIC). Scores on this single item measure range between 1 and 7 with higher scores reflecting greater impression of beneficial change.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rash, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (3):
- Canada (3):
  - Calgary Chronic Pain Centre, Calgary, Alberta
  - Jim Pattison Outpatient Care & Surgical Centre Pain Clinic (JPOCSC-PC), Surrey, British Columbia
  - Carbonear General Hospital, Carbonear, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified data (including data dictionaries) will be made available beginning 3-months after final follow-up data has been collected (anticipated September 2024) to researchers who provide a methodologically sound proposal for the purpose of achieving the aims of the approved proposal. Data sharing will be enacted with a data-transfer agreement between the sending and receiving institutions. Proposals should be directed to Joshua Rash (jarash@mun.ca)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3-months after final follow-up (anticipated September 2024). Data will remain available for 25-years.

REFERENCES:
- [Derived] Rash JA, Campbell TS, Cooper L, Flusk D, MacInnes A, Nasr-Esfahani M, Mekhael AA, Poulin PA, Robert M, Yi Y. Evaluating the efficacy of intranasal oxytocin on pain and function among individuals who experience chronic pain: a protocol for a multisite, placebo-controlled, blinded, sequential, within-subjects crossover trial. BMJ Open. 2021 Sep 23;11(9):e055039. doi: 10.1136/bmjopen-2021-055039. PMID 34556520